CLINICAL TRIAL: NCT00721370
Title: Near-Infrared Fluorescent Sentinel Lymph Node Mapping for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, John V. Frangioni, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2007P-000431
Record Dates: First submitted 2008-07-18; First posted 2008-07-24 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node mapping; breast cancer; near infrared imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients imaged using ICG:HSA and NIR imaging system
  Interventions: Device: NIR imaging system

INTERVENTIONS:
Device: NIR imaging system — Optical imaging parameter optimization (field-of-view, NIR excitation fluence rate, camera integration time) and system ergonomics.

SUMMARY:
Sentinel lymph node (SLN) mapping is the standard of care for the surgical staging of breast cancer. We propose a method of SLN mapping based on the use of invisible near-infrared fluorescent light that has significant advantages for both patient and surgeon. The present study is a 6-patient pilot study designed to optimize clinical workflow with the new imaging system.

DETAILED DESCRIPTION:
The standard of care in breast cancer surgery includes identification and assessment of the sentinel lymph node (SLN). At the present time, SLN mapping utilizes a gamma ray-emitting radiotracer and/or a blue dye. Radiotracers provide sensitive detection of SLNs, but require involvement of a nuclear medicine physician, vary widely in transit time depending on the agent employed, can be difficult to localize with a handheld gamma probe, and expose both patient and caregivers to ionizing radiation. Blue dyes, such as isosulfan blue, cannot be seen easily through skin and fat, but can aid in definitive identification of the SLN when the handheld gamma probe gives ambiguous results. Finally, the learning curve associated with expertise in the SLN procedure is quite long using currently available techniques.

In this 12-patient pilot study, we are testing a new intraoperative imaging system that we developed for image-guided surgery. The imaging system uses invisible, near-infrared (NIR) light to visualize lymphatic flow and to identify the SLN. The imaging system makes no contact with the patient and can display surgical anatomy simultaneously with NIR fluorescence.

All patients will receive the standard of care for SLN mapping, namely technetium-99m sulfur colloid lymphoscintigraphy. In addition, patients will be injected with indocyanine green (ICG) diluted in human serum albumin (HSA). ICG is already FDA approved for other indications and is used in this study at 400-fold to 2000-fold lower than the typical clinical dose. Dilution into HSA improves the brightness of ICG by over 3-fold, making it an excellent tracer for lymphatic flow.

The purpose of this pilot study is to determine whether the ergonomics of the imaging system interfere with typical clinical workflow during breast cancer surgery. A secondary goal is to optimize the imaging parameters (light levels, exposure time, etc.) associated with identification of the SLN.

ELIGIBILITY:
Inclusion Criteria:

* Women or men above the age of 21 who have biopsy-proven breast cancer, and who are undergoing sentinel lymph node mapping for staging and treatment of their disease.

Exclusion Criteria:

* Pregnant women,
* Significant renal, cardiac, or pulmonary disease,
* History of iodine allergy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Ergonomics and function of the imaging system - verify that the imaging system does not interfere with Sentinel Lymph Node mapping procedure and can be used safely by the surgeon. | Typical 1 hour clinical procedure

SECONDARY OUTCOMES:
Identify sentinel lymph nodes | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: John V Frangioni, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mieog JS, Troyan SL, Hutteman M, Donohoe KJ, van der Vorst JR, Stockdale A, Liefers GJ, Choi HS, Gibbs-Strauss SL, Putter H, Gioux S, Kuppen PJ, Ashitate Y, Lowik CW, Smit VT, Oketokoun R, Ngo LH, van de Velde CJ, Frangioni JV, Vahrmeijer AL. Toward optimization of imaging system and lymphatic tracer for near-infrared fluorescent sentinel lymph node mapping in breast cancer. Ann Surg Oncol. 2011 Sep;18(9):2483-91. doi: 10.1245/s10434-011-1566-x. Epub 2011 Mar 1. PMID 21360250
- See also: Website of the study principal investigator with detailed information about related work. — http://www.frangionilab.org